CLINICAL TRIAL: NCT03242083
Title: Evaluation de la Quality of Life in Secondary Atrophic Age-related Macular Degeneration
Brief Title: Evaluate the Quality of Life of Patients With AMD
Acronym: QUASAR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: KAUFFMANN PCA 2016
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary atrophic AMD
  Interventions: Other: quality of life questionnaire
- Secondary atrophic AMD
  Interventions: Other: quality of life questionnaire

INTERVENTIONS:
Other: quality of life questionnaire — quality of life questionnaire

SUMMARY:
Age-related macular degeneration (AMD) is a major cause of deep visual acuity loss. Because of progressive deterioration of the macula, patients with AMD complain about progressive visual problems that can impair their quality of life in the physical, mental and social domains. The principal objective principal of this study is to describe the evolution of quality of life between the diagnosis of secondary atrophic AMD and at 18 months after confirmation of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- For the 2 populations studied

* Persons who have given consent to take part
* Persons aged 50 years or older
* Willing and able to attend all of the scheduled visits and evaluations
* Macular atrophy or drusen measuring at least 125μm or multiple drusens measuring at least 63μm
* Atrophic AMD diagnosed on OCT and by autofluorescence and OCT angiography by 2 independent experienced assessors
* Diagnosed for less than 3 years
* MAVC score ≥ 19 letters (Equivalent Snellen ≥ 20/400), by using a scale at an initial distance of 4m

For patients with secondary atrophic AMD

• Secondary atrophic AMD, defined by persistent atrophic AMD at 1 year after the last injection of an anti-angiogenic agent, and at least 2 years after the first injection.

Exclusion Criteria:

General criteria

* Persons without national health insurance cover
* Physical or mental disability ruling out participation
* Inability to sign the written consent form, adults under guardianship
* Any participation in a study involving an experimental drug during the previous 3 months (dietary supplements are authorised).
* Adults under guardianship

General medical history

• Uncontrolled AHT

Ophthalmological history

* Severe non-proliferative or proliferative diabetic retinopathy
* Uncontrolled glaucoma (defined as an intra-ocular pressure greater than 30mmHg despite treatment with an anti-glaucoma agent) or a history of filtration surgery
* Corneal disease that could impair vision
* Monogenic macular dystrophy or toxic maculopathy
* History of uveitis
* Amblyopia of the eye concerned
* Intraocular surgery in the 3 months preceding inclusion
* History of cornea transplantation in the studied eye
* Treatment affecting vision: chloroquine and hydroxychloroquine, phenothiazine, tamoxifen, interferon (93), external radiotherapy of the face and neck

Ophthalmological examination

* Significant cataract (LOCS III grade of 5 or above, annexe 5.) (94)
* Active infection in either eye
* Central anterior serous or active retinopathy in either eye
* Choroid neo-vascularisation
* Active serous retinal detachment
* Refractive error less than -15D or more than +10D

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During an ophthalmology consultation, the clinician who has established the diagnosis of primary atrophic or secondarily atrophic AMD (defined in 1.1.2) proposes to the patient fulfilling the aforementioned eligibility criteria to participate in the study.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
responses to a quality of life questionnaire | Change compared with baseline score at month 6, month 12 and month 18

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France